#### **SUMMARY OF CHANGES – Consent**

NCI Protocol #: 10389 Local Protocol #:

**Protocol Version Date: 01/13/2022** 

**Protocol Title:** A Phase 1 Trial Combining WEE1 Inhibitor Adavosertib (AZD1775) with Radiation Therapy for Metastatic or Inoperable and Ineligible for Definitive Chemoradiation Esophageal and Gastroesophageal Junction Cancer

**Informed Consent Version Date:** 01/13/2022

#### **SUMMARY OF CHANGES – Consent**

| # | Section | Comments |
|---|---|---|
| 1. | Throughout | Updated protocol version in header |
| 2. | i | <ul> <li>Updated protocol version date.</li> <li>Updated informed consent version date</li> <li>Updated page numbers</li> </ul> |
| 3. | <u>Pg. 3</u> | Added "There is a risk of sepsis from taking AZD1775. Sepsis could be so severe that it could lead to death. The study team will discuss and document your decisions about sepsis with considerations for: 1) whether the physician has determined that therapy is beneficial and, if so, 2) whether or not you have chosen to continue the treatment." |
| 4. | <u>Pg. 17</u> | Added: signature line and date line for both participant and witness |

## **Research Study Informed Consent Document**

Study Title for Participants: Testing the addition of an anti-cancer drug, AZD1775, to radiation therapy for patients ineligible for definitive chemoradiation and who have metastatic or incurable esophageal and gastroesophageal junction cancers

Official Study Title for Internet Search on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>: Protocol 10389 A Phase 1 Trial Combining WEE1 Inhibitor Adavosertib (AZD1775) with Radiation Therapy for Metastatic or Inoperable and Ineligible for Definitive Chemoradiation Esophageal and Gastroesophageal Junction Cancer (NCT#TBD)

### **Overview and Key Information**

### What am I being asked to do?

We are asking you to take part in a research study. This study has public funding from the National Cancer Institute (NCI), part of the National Institutes of Health (NIH) in the United States Department of Health and Human Services. We do research studies to try to answer questions about how to prevent, diagnose, and treat diseases like cancer.

We are asking you to take part in this research study because you have esophageal cancer and gastroesophageal junction cancer that is not able to be treated with surgery or with chemotherapy and radiation therapy given at the same time or that has spread to other parts of your body.

### Taking part in this study is your choice.

You can choose to take part or you can choose not to take part in this study. You also can change your mind at any time. Whatever choice you make, you will not lose access to your medical care or give up any legal rights or benefits.

This document has important information to help you make your choice. Take time to read it. Talk to your doctor, family, or friends about the risks and benefits of taking part in the study. It's important that you have as much information as you need and that all your questions are answered. See the "Where can I get more information?" section for resources for more clinical trials and general cancer information.

## Why is this study being done?

This study is being done to answer the following question:

What is the highest dose of AZD1775 in combination with radiation therapy that can be safely and tolerably taken in patients with esophageal and gastroesophageal junction cancer that has

spread or is not removable by surgery, and is not able to be treated with standard chemotherapy and radiation therapy at the same time?

This is the first time this drug will be tested together in combination with radiation in adult patients without the addition of chemotherapy.

We are doing this study because we want to find out if this approach is better or worse than the usual approach for your esophageal and gastroesophageal junction cancer. The usual approach is defined as care most people get for esophageal and gastroesophageal junction cancer.

### What is the usual approach to my esophageal and gastroesophageal junction cancer?

The usual approach for patients who are not in a study is treatment with radiation alone or drugs which are FDA-approved. Sometimes, combinations of these treatments are used. For example, you may receive radiation therapy to treat the esophageal and gastroesophageal junction cancer and then receive chemotherapy after radiation. Your doctor can explain which treatment may be best for you. These treatments can reduce symptoms and may stop the tumor from growing for a few months or longer. Additional options include comfort care to help relieve symptoms.

### What are my choices if I decide not to take part in this study?

- You may choose to have the usual approach described above.
- You may choose to take part in a different research study, if one is available.
- You may choose not to be treated for cancer.
- You may choose to only get comfort care to help relieve your symptoms and not get treated for your cancer.

## What will happen if I decide to take part in this study?

If you decide to take part in this study, you will get the study drug, AZD1775, alone for one week, and then in combination with standard radiation therapy for up to three weeks (one cycle) of treatment, or until the side effects become too severe if you are in the dose escalation part of this study. If you are in the dose expansion part of this study, you will also get the study drug, AZD1775, for one week followed by 3 weeks of combination study drug and radiation therapy.

After you finish your treatment, your doctor and study team will watch you for side effects. They will check you three weeks after completing treatment with a clinic visit and then clinic visits will occur every 3 months for 2 years after treatment. After that, they will check you with clinic visits every 6 months for 3 years. This means you will keep seeing your doctor for a total of 5 years after treatment. If you have persistent side effects, you will be required to meet with your study team more frequently.

### What are the risks and benefits of taking part in this study?

There are both risks and benefits to taking part in this study. It is important for you to think carefully about these as you make your decision.

#### Risks

We want to make sure you know about a few key risks right now. We give you more information in the "What risks can I expect from taking part in this study?" section.

If you choose to take part in this study, there is a risk that the study drug may not be as good as the usual approach alone at shrinking or stabilizing your cancer.

There is also a risk that you could have side effects from the study drug. These side effects may be worse and may be different than you would get with the usual approach for your cancer.

Some of the most common side effects that the study doctors know about are:

- Painful swallowing
- Diarrhea
- Nausea
- Vomiting
- Tiredness

Combining the study drug with standard radiation can result in greater similar side effects of those currently experienced by either the drug or by radiation alone.

While taking the study drug, AZD1775, there is a risk of developing an infection that can travel by blood and infect other parts of your body. The study team will discuss and document your decisions about this and other risk factors. The study team will discuss and document whether the physician has determined that therapy is beneficial and if so, whether or not you choose to continue the treatment.

There may be some risks that the study doctors do not yet know about.

#### **Benefits**

There is some evidence in living human cells that adding AZD1775 to the usual approach can stabilize cancer for longer than the usual approach alone. However, we do not know if this will happen in people. It is unlikely that this AZD1775 will help you live longer than the usual approach alone. This study may help the study doctors learn things that may help other people in the future.

## If I decide to take part in this study, can I stop later?

Yes, you can decide to stop taking part in the study at any time.

If you decide to stop, let your study doctor know as soon as possible. It's important that you stop safely. If you stop, you can decide if you want to keep letting the study doctor know how you are doing.

Your study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

## Are there other reasons why I might stop being in the study?

Yes. The study doctor may take you off the study if:

- Your health changes and the study is no longer in your best interest.
- New information becomes available and the study is no longer in your best interest.
- You do not follow the study rules.
- For women: You become pregnant while on the study.
- The study is stopped by Institutional Review Board (IRB), Food and Drug Administration (FDA), or study sponsor (NCI). The study sponsor is the organization who oversees the study.

It is important that you understand the information in the informed consent before making your decision. Please read, or have someone read to you, the rest of this document. If there is anything you don't understand, be sure to ask your study doctor or nurse.

### What is the purpose of this study?

The purpose of this study is to test the safety and tolerability (side effects) of adding a study drug called AZD1775 at different doses along with standard radiation treatment. This study tests different doses of the study drug when given with radiation at various times to see which dose is safer and more tolerable for people. There will be about 33 people taking part in this study. "Dose" is defined as the amount of drug you get (such as 150 mg). We want to find out what effects (good or bad) the drug has on people, if any. In addition, another objective of the study is to perform genetic testing on your tumor tissue to determine if certain genetic changes in the tumor help predict who will respond to the drug. Also, we will look for specific changes in the tumor which occur following treatment which indicate response to the drug.

## What are the study groups?

There are two parts in this study, a dose escalation part and a dose expansion part. Your doctor will tell you which part you are in.

In the dose escalation part of this study, different people will get different doses of the study drug AZD1775.

The first two people taking part in this study will get the first dose. If the drug does not cause serious side effects, the next group of people in the study will get a higher dose. The study doctor will watch each group carefully as they increase the dose. The doses will continue to increase for every new group until reaching the highest planned dose or there are serious side

effects that require the dose to be lower. If the latter occurs, dose escalation is stopped and patients will be treated at the lower dose.

In the dose expansion part of this study, the highest dose with manageable side effects will be given to 12 more people. This will help study doctors better understand the side effects that may happen with this drug.

Treatment schedule: In the dose escalation and dose expansion part of this study, you will get AZD1775 as a capsule you take by mouth alone for two to five days per week for one week (Week -1). Then, you will take the AZD1775 by mouth 2-3 hours before radiation therapy two to five days per week during the first and third weeks of radiation therapy. Your doctor will tell you how often you should take the AZD1775. Radiation therapy will be given five days per week for three weeks total. See the study calendar for more information.

This drug, either alone or in combination with radiation, is not approved by the FDA for treatment of your disease.

### What exams, tests, and procedures are involved in this study?

Before you begin the study, your doctor will review the results of your exams, tests, and procedures. This helps your doctor decide if it is safe for you to take part in the study. If you join the study, you will have more exams, tests, and procedures to closely monitor your safety and health. Most of these are included in the usual care you would get even if you were not in a study.

Listed below are exams, tests, and procedures that need to be done as part of this study to monitor your safety and health, but may not be included in the usual care. We will use them to carefully follow the effects of the study treatment, including preventing and managing side effects.

These exams, tests, and procedures to monitor your safety and health include:

- Blood counts done weekly during treatment.
- Physical exams done weekly during treatment.

This study will use genetic tests that may identify changes in the genes in your DNA. Your genes carry information about you and your family, from the color of your eyes to health conditions for which you may be at risk, such as certain kinds of cancer.

Finding these changes would not affect your treatment in this study. However, they could affect your health in other ways. If the changes in your genes were inherited, the changes could also affect the health of your family members. Results from genetic testing will not be a part of your medical records, unless the results are confirmed by additional testing that you agreed to. See "Who will see my medical information?" for laws and risks in protecting your genetic information.

Some exams, tests, and procedures are a necessary part of the research study, but would not be included in usual care. Listed below are procedures that will be done for research purposes only.

Your study doctor will need to use some of the tissue left over from your biopsy when you were diagnosed with cancer. This sample is a required part of the study. This sample will be used to predict if this treatment will work for your type of cancer. You or your study doctor will get the results of this testing.

If there is not enough tissue left over from your biopsy, your study doctor will need to do a mandatory biopsy to get this tissue. This biopsy will be collected before you begin taking the study drug. The study biopsy takes small pieces of cancer tissue from your body. This is like the biopsy you had that helped diagnose your cancer. This sample will be used to predict if this treatment will work for your type of cancer.

If you are in the dose expansion cohort, you will need to have two mandatory biopsies for the study. The study biopsy takes small pieces of cancer tissue from your body. This is like the biopsy you had that helped diagnose your cancer. The first biopsy will be done before you begin the study drug. If a tumor tissue sample cannot be obtained by biopsy or by using left over tissue, your study doctor will let you know if you are still able to participate in the study. An additional mandatory biopsy will be collected on the fourth or fifth day of treatment.

Mandatory blood samples will also be taken for the study. The blood sample will be collected before you begin the study drug. The blood samples will be used to help identify genetic changes in your tumor which can be used to predict response to the drug.

A patient study calendar is attached at the end of this document. It shows how often these procedures will be done.

## What risks can I expect from taking part in this study?

#### **General Risks**

If you choose to take part in this study, there is a risk that the study drug may not be as good as the usual approach for your cancer or condition at shrinking or stabilizing your cancer.

You also may have the following discomforts:

- Spend more time in the hospital or doctor's office.
- Be asked sensitive or private questions about things you normally do not discuss.
- May not be able to take part in future studies.

The study drug in combination with radiation therapy used in this study could be very harmful to an unborn or newborn baby. There may be some risks that doctors do not yet know about. It is very important that you check with your study doctor about what types of birth control or pregnancy prevention to use during the study and for 1 month after you have completed the study.

This study will use a sample of your tissue. Generally, your hospital will keep some of your tissue. This tissue may be used to help treat your cancer in the future. Because this study will need to use some of this tissue, there is a small risk that it could be used up.

#### **Genetic Testing Risks**

The genetic test used in this study will test your tumor and normal tissue to identify changes in genes that help repair your DNA. Changes found in your normal tissue may be passed down in families. For example, these genetic changes may be passed down to your children in the same way that eye and hair color are passed down.

Genetic tests of normal tissue can reveal information about you and also about your relatives. Your doctor will talk with you about what the tests results may mean for you and your family. He or she also may suggest you talk with a genetics counselor to learn more. You or your insurance plan would have to pay for visits to a genetic counselor.

#### **Biopsy Risks**

Common side effects of a biopsy are a small amount of bleeding at the time of the procedure, bruising, and pain at the biopsy site. Pain can be treated with regular pain medications. Rarely, an infection, significant bleeding, or collapsing of the lung can occur. You may sign a separate consent form for the study biopsy that describes the risks in more detail.

#### **Blood Draw Risks**

Some of the risks from drawing blood from your arm may include pain, bruising, light-headedness, and rarely, infection. For most people, needle punctures to get blood samples do not cause any serious harm. Let your study doctor know of any questions you have about possible side effects. You can ask the study doctor questions about side effects at any time.

#### **Side Effect Risks**

The study drug and radiation therapy used in this study may affect how different parts of your body work such as your liver, kidneys, heart, lungs, and blood. The study doctor will test your blood and let you know if changes occur that may affect your health.

There is also a risk that you could have other side effects from the study drug and radiation therapy.

Please note that the study goal is to find a dose of the study drug where there is a one in four chance that a severe toxicity occurs in the first 28 days of treatment or subsequent 3 week follow-up period.

Here are important things to know about side effects:

- 1. The study doctors do not know who will or will not have side effects.
- 2. Some side effects may go away soon, some may last a long time, and some may never go away.
- 3. Some side effects may make it hard for you to have children.
- 4. Some side effects may be mild. Other side effects may be very serious and even result in death.

You can ask your study doctor questions about side effects at any time. Here are important ways to make side effects less of a problem:

- If you notice or feel anything different, tell your study doctor. He or she can check to see if it is a side effect.
- Your study doctor will work with you to treat your side effects.
- Your study doctor may adjust the study drugs to try to reduce side effects.

You should notify your doctor immediately at the first sign of poorly formed or loose stools or an increased frequency of bowel movements. Loperamide (Imodium) should be kept on hand and should be taken as recommended by your doctor.

#### **Drug Risks**

The tables below show the most common and most serious side effects doctors know about. Keep in mind that there might be other side effects doctors do not yet know about. If important new side effects are found, the study doctor will discuss these with you.

#### **Possible Side Effects of AZD1775**

(Table Version Date: April 27, 2020)

#### **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving AZD1775 (adavosertib), more than 20 and up to 100 may have:

- Diarrhea, nausea, vomiting
- Tiredness

#### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving AZD1775 (adavosertib), from 4 to 20 may have:

- Anemia which may require blood transfusion
- Pain
- Constipation, heartburn
- Sores in the mouth which may cause difficulty swallowing
- Swelling of the body
- Fever
- Infection, especially when white blood cell count is low
- Bruising, bleeding
- Weight loss, loss of appetite
- Dehydration
- Dizziness, headache
- Difficulty sleeping
- Cough, shortness of breath
- Rash

#### RARE, AND SERIOUS

In 100 people receiving AZD1775 (adavosertib), 3 or fewer may have:

- Abnormal heartbeat
- Bleeding from multiple sites
- Internal bleeding which may cause black tarry stool, blood in vomit
- Damage to the liver
- Change in the heart rhythm
- Bleeding in the brain which may cause confusion

#### **Additional Drug Risks**

The study drug could interact with other drugs. While being in the study, you should avoid certain medications that are strong inducers/inhibitors or substrates of CYP 3A4, 2C19, OATP1B1, OATP1B3, MATE1, MATE2K, P-gp, and BCRP. Your study doctor will give you a drug information handout and wallet card that lists these possible interactions. Share this information with your family members, caregivers, other health care providers, and pharmacists.

Rarely, there are problems getting enough supplies of the study drug. If that happens, your doctor will talk with you about your options.

#### **Possible Side Effects of Radiation Therapy**

#### **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving radiation therapy, 20 to 100 may have:

- Reddening, tanning, or peeling of the skin
- Mild pain
- Hair loss
- Tiredness
- Diarrhea, nausea
- Anemia, which may require transfusion
- Infection, especially when white blood cell count is low

#### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving radiation therapy, 4 to 20 may have:

- Thickening and numbness of the skin
- Sores or ulcers on the skin or near the cancer location
- Permanent hair loss
- Bleeding from the skin
- Sores in mouth which may cause difficulty swallowing

#### RARE, AND SERIOUS

In 100 people receiving radiation therapy, 3 or fewer may have:

- Damage to internal organs
- Abnormal opening in internal organs which may cause pain and bleeding

## What are my responsibilities in this study?

If you choose to take part in this study you will need to:

- Keep your study appointments.
- Tell your doctor about:
  - o all medications and supplements you are taking
  - o any side effects
  - o any doctors' visits or hospital stays outside of this study
  - o if you have been or are currently in another research study.
- Write down in your medication diary when you take the study drug at home.

**For women:** Do not get pregnant or breastfeed while taking part in this study. **For men:** Do not father a baby while taking part in this study. **For all:** Tell your study doctor right away if you think that you or your partner have become pregnant during the study or within 1 month after your last dose of study treatment.

## What are the costs of taking part in this study?

You and/or your insurance plan will need to pay for the costs of medical care you get as part of the study, just as you would if you were getting the usual care for your cancer. This includes:

- the costs of tests, exams, procedures, and drugs that you get during the study to monitor your safety, and prevent and treat side effects.
- your insurance co-pays and deductibles.
- biopsy specimen collection taken prior to starting treatment if there is not enough tissue left over from the biopsy which was performed when you were diagnosed with cancer

Talk to your insurance provider and make sure that you understand what your insurance pays for and what it doesn't pay for if you take part in this clinical trial. Also, find out if you need approval from your plan before you can take part in the study.

Ask your doctor or nurse for help finding the right person to talk to if you are unsure which costs will be billed to you or your insurance provider.

You and/or your insurance provider will not have to pay for exams, tests, and procedures done for research purposes only or that are covered by the study. These include:

- The blood specimen collected prior to treatment for research purposes
- The examination and biopsy of your esophagus tumor performed prior to starting treatment and on the fourth or fifth day of treatment (week -1), if you are part of the expansion cohort.

You or your insurance provider will not have to pay for the AZD1775 while you take part in this study.

Taking part in this study may mean that you need to make more visits to the clinic or hospital than if you were getting the usual approach to treat your cancer. You may:

- Have more travel costs.
- Need to take more time off work.
- Have other additional personal costs.

You will not be paid for taking part in this study. The research may lead to new tests, drugs, or other products for sale. If it does, you will not get any payment.

## What happens if I am injured because I took part in this study?

If you are injured as a result of taking part in this study and need medical treatment, please talk with your study doctor right away about your treatment options. The study sponsors will not pay for medical treatment for injury. Your insurance company may not be willing to pay for a study-related injury. Ask them if they will pay. If you do not have insurance, then you would need to pay for these medical costs.

Page 12 of 19

If you feel this injury was caused by medical error on the part of the study doctors or others involved in the study, you have the legal right to seek payment, even though you are in a study. Agreeing to take part in this study does not mean you give up these rights.

### Who will see my medical information?

Your privacy is very important to us. The study doctors will make every effort to protect it. The study doctors have a privacy permit to help protect your records if there is a court case. However, some of your medical information may be given out if required by law. If this should happen, the study doctors will do their best to make sure that any information that goes out to others will not identify who you are.

Some of your health information, such as your response to cancer treatment, results of study tests, and medicines you took, will be kept by the study sponsor in a central research database. However, your name and contact information will not be put in the database. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used.

There are organizations that may look at or receive copies of some of the information in your study records. Your health information in the research database also may be shared with these organizations. They must keep your information private, unless required by law to give it to another group.

Some of these organizations are:

- The study sponsor and any company supporting the study agent now or in the future. This would include any organization helping the company with the study.
- The NCI Central IRB, which is a group of people who review the research with the goal of protecting the people who take part in the study.
- The FDA and the groups it works with to review research.
- The NCI and the groups it works with to review research.

In addition to storing data in the study database, data from studies that are publicly funded may also be shared broadly for future research with protections for your privacy. The goal of this data sharing is to make more research possible that may improve people's health. Your study records may be stored and shared for future use in public databases. However, your name and other personal information will not be used.

Some types of future research may include looking at your information and information from other patients to see who had side effects across many studies or comparing new study data with older study data. However, right now we don't know what research may be done in the future using your information. This means that:

• You will not be asked if you agree to take part in the specific future research studies using your health information.

- You and your study doctor will not be told when or what type of research will be done.
- You will not get reports or other information about any research that is done using your information.

There are laws that protect your genetic information. However, there is a risk that someone could get access to your genetic information and identify you by name. In some cases, employers could use your genetic information to decide whether to hire or fire you. The study doctors believe the risk of this happening is very small. However, the risk may increase in the future as people find new ways of tracing information. For more information about the laws that protect you, ask your study doctor.

### Where can I get more information?

You may visit the NCI web site at http://cancer.gov/ for more information about studies or general information about cancer. You may also call the NCI Cancer Information Service to get the same information at: 1-800-4-CANCER (1-800-422-6237).

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

You can talk to the study doctor about any questions or concerns you have about this study or to report side effects or injuries. Contact the study doctor (\*insert name of study doctor[s]\*) at (\*insert telephone number, and email address if appropriate\*).

For questions about your rights while in this study, call the (\*insert name of organization or center\*) Institutional Review Board at (\*insert telephone number\*).

## Optional studies that you can choose to take part in

This part of the consent form is about optional studies that you can choose to take part in. They are separate from the main study described above. These optional studies will not benefit your health. The researchers leading this optional study hope the results will help other people with cancer in the future. The results will not be added to your medical records and you or your study doctor will not know the results.

Taking part in this optional study is your choice. You can still take part in the main study even if you say "no" to this study. There is no penalty for saying "no." You and your insurance company will not be billed for this optional study. If you sign up for, but cannot complete this study for any reason, you can still take part in the main study.

Circle your choice of "yes" or "no" for the following study.

## Optional sample collections for storage for possible future studies

Researchers are trying to learn more about cancer and other health problems using blood and tissue samples from people who take part in clinical trials. By studying these samples, researchers hope to find new ways to prevent, detect, treat, or cure diseases.

Some of these studies may be about how genes affect health and disease. Other studies may look at how genes affect a person's response to treatment. Genes carry information about traits that are found in you and your family. Examples of traits are the color of your eyes, having curly or straight hair, and certain health conditions that are passed down in families. Some of the studies may lead to new products, such as drugs or tests for diseases.

If you are in the dose expansion group and choose to take part in this optional study, a sample of tissue from your biopsy prior to starting the drug and the repeat biopsy obtained during the first week of drug will be collected and stored. Storing samples for future studies is called "biobanking." The biobank is being run by ETCTN Biorepository and is supported by the NCI. Also, any health-related information, such as your response to cancer treatment, results of study tests, and medicines you took, will be stored for future use. This is a publicly funded study. Samples from publicly funded studies are required to be shared as broadly as possible. However, we will protect your privacy. The goal of this is to make more research possible that may improve people's health.

The biobank is a public research resource. It has controlled access. This means that researchers who want to get samples and data from it must submit a specific research request. The request identifies who they are and what their planned research project is. Before getting the samples and data, the researchers must agree to keep the data private, only use it for their planned research project, and never use it to try to identify you.

Right now, we don't know what research may be done in the future using your tissue samples. This means that:

- You will not be asked if you agree to take part in the future research studies.
- You and your study doctor will not be told when or what type of research will be done.
- You will not get reports or other information about any research that is done using your samples.

Unknown future research studies may include sequencing of all or part of your DNA. This is called genomic sequencing. Sequencing allows researchers to identify your genetic code. Changes in your genetic code may just be in your tumor tissue. These are called somatic changes. Changes may also be in your normal tissue and passed down through your family. For example, these genetic changes may be passed down to your children in the same way that eye and hair color are passed down. These are called germline changes.

If only tumor tissue is sequenced, we will not know if a genetic change in your tumor is also in your normal tissue. This is why sometimes both normal tissue and tumor tissue are sequenced. This helps researchers understand if a genetic change happened only in your cancer tissue, or in your normal tissue as well.

### What is involved in this optional sample collection?

If you agree to take part, here is what will happen next:

- 1. If you are in the dose expansion group, an extra sample of tissue will be collected during the biopsy prior to treatment and again on Day 4 or 5 of Week -1. For the biopsy procedure, the study doctor will take pieces of your tumor during a procedure to evaluate the esophageal and gastroesophageal junction tumor. This process may be repeated several times in the same procedure in order to get enough tissue.
- 2. Your samples will be stored in the biobank. There is no limit on the length of time we will keep your samples and research information. The samples will be kept until they are used for research or destroyed.
- 3. Researchers can only get samples from the biobank after their research has been approved by experts. Researchers will not be given your name or contact information.
- 4. Some of your genetic and health information may be placed in central databases for researchers to use. The databases will not include your name or contact information.

### What are the risks in this optional sample collection?

- The most common risks related to a biopsy are a small amount of bleeding at the time of the procedure, bruising, and pain at the biopsy site. Pain can be treated with regular pain medications. Rarely, an infection, significant bleeding, or collapsing of the lung can occur. The most common risks related to drawing blood from your arm are brief pain and maybe a bruise.
- Generally, hospitals will keep some of your tissue. This tissue may be used to help treat your cancer in the future. There is a small risk that when this tissue sample is submitted to the biobank for this optional sample collection, your tissue could be used up.
- Your medical and genetic information is unique to you. There is a risk that someone outside of the research study could get access to your study records or trace information in a database back to you. They could use that information in a way that could harm you. Researchers believe the chance that someone could access and misuse your information is very small. However, the risk may increase in the future as people find new ways of tracing information.
- In some cases, this information could be used to make it harder for you to get or keep a job and get or keep health insurance. There are laws against the misuse of genetic information, but they may not give full protection. For more information about the laws that protect you, ask your study doctor or visit: https://www.genome.gov/10002328/

#### How will information about me be kept private?

Your privacy is very important to the study researchers and biobank. They will make every effort to protect it. Here are just a few of the steps they will take:

1. They will remove identifiers, such as your initials, from your sample and information. They will replace them with a code number. There will be a master list linking the code numbers to names, but they will keep it separate from the samples and information. Only

your study doctor and a few study researchers will have access to the master list linking the code numbers to names. The biobank and the genomic sequencing laboratory will receive your samples with the following information only: your sample code number; your age, race/ethnicity, and gender; your type of cancer; any previous treatments you received for your cancer; and the treatment you will receive for this current study.

- 2. Researchers who study your samples and information will not know who you are. They also must agree that they will not try to find out who you are. The researchers must be trained in the handling of private information. Any researcher who wants to study your stored samples and genetic information must apply and be approved to do so.
- 3. Your personal information will not be given to anyone unless it is required by law.
- 4. If research results are published, your name and other personal information will not be used.

#### What are the benefits to taking part in this optional sample collection?

You will not benefit from taking part.

The researchers, using the samples from you and others, might make discoveries that could help people in the future.

#### Are there any costs or payments to this optional sample collection?

There are no costs to you or your insurance for exams, tests, and procedures done for research purposes only; these include the biopsy, blood draw, DNA/RNA sequencing, and biobanking of your specimen(s). You will not be paid for taking part in this study. The research may lead to new tests, drugs, or other products for sale. If it does, you will not get any payment.

#### What if I change my mind about this optional sample collection?

If you decide you no longer want your samples to be used, you can call the study doctor, (\*insert name of study doctor[s]\*) at (\*insert telephone number, and email address if appropriate\*), who will let the biobank know. Then, any sample that remains in the biobank will be destroyed or returned to your study doctor. This will not apply to any samples or related health information that have already been given to or used by researchers.

#### What if I have questions about this optional sample collection?

If you have questions about the use of your samples for research, contact the study doctor, (\*insert name of study doctor[s]\*) at (\*insert telephone number, and email address if appropriate\*).

Please circle your answer below to show if you would or would not like to take part in each optional study:

#### Samples for unknown future studies:

| I agree that my sar | mples and | related hea | ılth informa | ıtion may b | oe kept ir | n a biobank : | for use in | future |
|---|---|---|---|---|---|---|---|---|
| health research. | | | | | | | | |

YES NO

#### **Contact for Future Research**

I agree that my study doctor, or someone on the study team, may contact me or my doctor to see if I wish to participate in other research in the future.

YES NO

Participant's signature:

This is the end of the section about optional studies.

## My signature agreeing to take part in the study

I have read this consent form or had it read to me. I have discussed it with the study doctor and my questions have been answered. I will be given a signed and dated copy of this form. I agree to take part in the main study. I also agree to take part in any additional studies where I circled "yes".

| | _ |
|---------------------------------------------------------------|-------|
| Date of signature: | |
| Signature of person(s) conducting the informed conliscussion: | ısent |
| Date of signature: | |

# **Patient Study Calendar**

| | Pre-Treatment | | | | During | g Treatmo | ent | Follow-Up | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | ≤12<br>month<br>s prior<br>to<br>study<br>entry | ≤28 days prior to study entry | ≤14<br>days<br>prior<br>to<br>study<br>entry | Wk<br>-1 | Wk<br>1 | Wk<br>2 | Wk<br>3 | Wk<br>6 | Every 3 months<br>(+/- 1 month) for<br>first 2 years | Every 6 months (+/-1 month) for years 2-5 |
| AZD1775 <sup>a</sup> | | | | X | X | | X | | | |
| Informed consent | | X | | | | | | | | |
| Medical history and physical exam | | | X | | X | X | X | X | X | X |
| Vital signs | | | X | | X | X | X | X | X | X |
| Weight and an assessment<br>of how well you perform<br>everyday tasks and<br>activities | | | X | | X | X | X | X | X | X |
| Blood draws for complete<br>blood count and general<br>health status | | | X | | X | X | X | X | X | X |
| EKG | | X | | As indicated by your doctor | | | | | | |
| Blood or urine collection<br>for pregnancy test (for<br>women of childbearing<br>potential) | | X | | Performed on Day 1 | | | | | | |
| Side effect evaluation | | | | X | | | | X | | |
| Medical imaging scans for tumor measurements | | X | | | | | | | | |
| Test to examine your<br>throat, stomach, and<br>intestines, along with a<br>biopsy | X | | X<br>(expa<br>nsion<br>cohort<br>only) | Performed<br>on Day 4<br>or 5<br>(expansion<br>cohort<br>only) | | | | | | |
| Radiation therapy <sup>b</sup> | | | | | X | X | X | | | |
| Assessment of how well<br>you are able to swallow<br>(expansion cohort only) | | | X | | | | | X | X | X |
| Tumor tissue collection for research purposes | | X <sup>c</sup> | | | | | | | | |
| Mandatory Tumor tissue<br>collection for research<br>purposes (expansion<br>cohort only) | | | X | Performed<br>on Day 4<br>or 5 | | | | | | |

| | Pre-Treatment | | | During Treatment | | | | | Follow-Up | |
|---|---|---|---|---|---|---|---|---|---|---|
| | ≤12<br>month<br>s prior<br>to<br>study<br>entry | ≤28 days prior to study entry | ≤14<br>days<br>prior<br>to<br>study<br>entry | Wk<br>-1 | Wk<br>1 | Wk<br>2 | Wk<br>3 | Wk<br>6 | Every 3 months<br>(+/- 1 month) for<br>first 2 years | Every 6 months (+/-1 month) for years 2-5 |
| Optional Tumor tissue<br>collection for research<br>purposes (expansion<br>cohort only) | | | X | Performed<br>on Day 4<br>or 5 | | | | | | |
| Mandatory Blood<br>collection for research<br>purposes | | X | | | | | | | | |

a: Dose as assigned, 2-3 hours prior to radiation therapy during the first and third weeks of radiation therapy.

b: Delivered five days per week.

c: If tumor tissue from your previous biopsies is not available, this biopsy is mandatory.